CLINICAL TRIAL: NCT00018681
Title: Regulation of Human Intestinal Bile Acid Transport in Health and Disease
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: GAST-005-98S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study investigates distribution and regulation of bile acid transport in the human intestine.

ELIGIBILITY:
Veterans, healthy, scheduled for screening colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-04; Study Completion 2002-01

CONTACTS AND LOCATIONS:
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States